CLINICAL TRIAL: NCT04825015
Title: Hemodynamic Monitoring in Liver Transplant With VEnaRt Cardiac Output Versus Swan-Ganz Catheter VERO Study
Brief Title: Hemodynamic Monitoring in Liver Transplant With VEnaRt Cardiac Output Versus Swan-Ganz Catheter (VERO Study)
Acronym: VERO
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: CEUR-2020-OS-299
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Output, Low; Liver Transplant; Complications
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- OLTx: Liver insufficiency patients undergoing transplantation surgery
  Interventions: Device: VEnaRt Cardiac Output

INTERVENTIONS:
Device: VEnaRt Cardiac Output — Every patient is monitored during liver transplantation with VEnaRt Cardiac Output versus Swan-Ganz Catheter

SUMMARY:
The Swan-Ganz catheter is the gold standard to measure cardiac output during liver transplantation surgery. This is an invasive hemodynamic monitoring system.

The VenArt Cardiac Output (Mespere LifeSciences, Waterloo, Canada) is a new, innovative and non-invasive device that permits hemodynamic monitoring.

With a software based on Fick's principle it is able to calculate cardiac output, cardiac index and continuous cardiac output.

The hypothesis of this study is to investigate the precision and accuracy of this method versus the standard of care during liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation patients

Exclusion Criteria:

* age < 18 years old
* combined liver-kidney transplant
* liver transplant for acute insufficiency
* no consent of the patient

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients undergoing liver transplant at our institution
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Precision of VenArt Cardiac Output cardiac output, cardiac index and continuous cardiac output measures | During surgery
  Evaluate the precision of VenArt Cardiac Output cardiac output, cardiac index and continuous cardiac output versus the pulmonary catheter in patients undergoing liver transplantation
Accuracy of VenArt Cardiac Output cardiac output, cardiac index and continuous cardiac output measures | During surgery
  Evaluate the accuracy of VenArt Cardiac Output cardiac output, cardiac index and continuous cardiac output versus the pulmonary catheter in patients undergoing liver transplantation

SECONDARY OUTCOMES:
Correlation | During surgery
  Analyze the VenArt Cardiac Output and Swan-Ganz catheter statistical correlation of cardiac output and cardiac index measures
Concordance | During surgery
  Analyze the VenArt Cardiac Output and Swan-Ganz catheter statistical concordance of cardiac output and cardiac index measures
Time of device positioning | During surgery
  Evaluate the time necessary to position the VenArt Cardiac Output and Swan-Ganz catheter
Device positioning complications | During surgery
  Evaluate the complication during the VenArt Cardiac Output and Swan-Ganz catheter positioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Wolf AM. Pulmonary artery catheter: rest in peace? Not just quite yet.. Liver Transpl. 2008 Jul;14(7):917-8. doi: 10.1002/lt.21543. No abstract available. PMID 18581507
- [Background] Rudnick MR, Marchi LD, Plotkin JS. Hemodynamic monitoring during liver transplantation: A state of the art review. World J Hepatol. 2015 Jun 8;7(10):1302-11. doi: 10.4254/wjh.v7.i10.1302. PMID 26052376
- [Background] Cecconi M, Dawson D, Casaretti R, Grounds RM, Rhodes A. A prospective study of the accuracy and precision of continuous cardiac output monitoring devices as compared to intermittent thermodilution. Minerva Anestesiol. 2010 Dec;76(12):1010-7. Epub 2010 Jul 16. PMID 20634793
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Weinbroum AA, Biderman P, Soffer D, Klausner JM, Szold O. Reliability of cardiac output calculation by the fick principle and central venous oxygen saturation in emergency conditions. J Clin Monit Comput. 2008 Oct;22(5):361-6. doi: 10.1007/s10877-008-9143-y. Epub 2008 Oct 23. PMID 18946716
- [Background] Critchley LA, Critchley JA. A meta-analysis of studies using bias and precision statistics to compare cardiac output measurement techniques. J Clin Monit Comput. 1999 Feb;15(2):85-91. doi: 10.1023/a:1009982611386. PMID 12578081
- [Background] Critchley LA, Lee A, Ho AM. A critical review of the ability of continuous cardiac output monitors to measure trends in cardiac output. Anesth Analg. 2010 Nov;111(5):1180-92. doi: 10.1213/ANE.0b013e3181f08a5b. Epub 2010 Aug 24. PMID 20736431
- [Background] Vetrugno L, Bignami E, Barbariol F, Langiano N, De Lorenzo F, Matellon C, Menegoz G, Della Rocca G. Cardiac output measurement in liver transplantation patients using pulmonary and transpulmonary thermodilution: a comparative study. J Clin Monit Comput. 2019 Apr;33(2):223-231. doi: 10.1007/s10877-018-0149-9. Epub 2018 May 3. PMID 29725794